CLINICAL TRIAL: NCT05330975
Title: A Phase 3 Randomized, Observer-Blind, Study to Evaluate Safety, Tolerability, and Immunogenicity of mRNA-1345, an mRNA Vaccine Targeting Respiratory Syncytial Virus (RSV), When Given Alone or Coadministered With a Seasonal Influenza Vaccine or SARS-CoV-2 Vaccine and When Given as an Open-label Boost at 1 Year Following a Primary Dose in Adults ≥ 50 Years of Age
Brief Title: A Study of mRNA-1345 Vaccine Targeting Respiratory Syncytial Virus (RSV) in Adults ≥50 Years of Age
Acronym: RSVictory
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1345-P302
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Syncytial Virus
Keywords: Viral Diseases; Messenger RNA; Moderna; mRNA-1345; Respiratory syncytial virus; Safety; Vaccines; SARS-CoV-2
MeSH Terms: conditions — Virus Diseases | interventions — mRNA-1345 respiratory syncytial virus vaccine; mRNA-1273.214 COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Parts A and B are randomized, observer blind studies and Part C is a single-arm, open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part A: mRNA-1345 + Placebo (Experimental): Single injection of mRNA-1345 and placebo, administered intramuscularly (IM), one in each arm on Day 1.
  Interventions: Biological: Placebo; Biological: mRNA-1345
- Part A: mRNA-1345 + Afluria® Quadrivalent (Experimental): Single injection of mRNA-1345 and Afluria® quadrivalent, administered IM, one in each arm on Day 1.
  Interventions: Biological: mRNA-1345; Biological: Afluria® Quadrivalent
- Part A: Afluria® Quadrivalent + Placebo (Active Comparator): Single injection of Afluria® quadrivalent and placebo, administered IM, one in each arm on Day 1.
  Interventions: Biological: Placebo; Biological: Afluria® Quadrivalent
- Part B: mRNA-1345 + Placebo (Experimental): Single injection of mRNA-1345 and placebo, administered IM, one in each arm on Day 1. An additional injection of mRNA-1273.214, administered on Day 29.
  Interventions: Biological: Placebo; Biological: mRNA-1345; Biological: mRNA-1273.214
- Part B: mRNA-1345 + mRNA-1273.214 (Experimental): Single injection of mRNA-1345 and mRNA-1273.214, administered IM, one in each arm on Day 1. An additional injection of placebo administered on Day 29.
  Interventions: Biological: Placebo; Biological: mRNA-1345; Biological: mRNA-1273.214
- Part B: mRNA-1273.214 + Placebo (Active Comparator): Single injection of mRNA-1273.214 and placebo, administered IM, one in each arm on Day 1. An additional injection of placebo administered on Day 29.
  Interventions: Biological: Placebo; Biological: mRNA-1273.214
- Part C: mRNA-1345 (Experimental): Single injection of mRNA-1345 administered IM on BD Day 1.
  Interventions: Biological: mRNA-1345

INTERVENTIONS:
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Part A: Afluria® Quadrivalent + Placebo; Part A: mRNA-1345 + Placebo; Part B: mRNA-1273.214 + Placebo; Part B: mRNA-1345 + Placebo; Part B: mRNA-1345 + mRNA-1273.214
Biological: mRNA-1345 — Sterile liquid for injection
  Arms: Part A: mRNA-1345 + Afluria® Quadrivalent; Part A: mRNA-1345 + Placebo; Part B: mRNA-1345 + Placebo; Part B: mRNA-1345 + mRNA-1273.214; Part C: mRNA-1345
Biological: Afluria® Quadrivalent — single-dose, pre-filled syringe for injection
  Arms: Part A: Afluria® Quadrivalent + Placebo; Part A: mRNA-1345 + Afluria® Quadrivalent
Biological: mRNA-1273.214 — Sterile liquid for injection
  Arms: Part B: mRNA-1273.214 + Placebo; Part B: mRNA-1345 + Placebo; Part B: mRNA-1345 + mRNA-1273.214

SUMMARY:
The main purposes of Part A of this study are to evaluate the safety, tolerability, and immunogenicity of mRNA-1345 coadministered with a seasonal influenza vaccine (Afluria® Quadrivalent); to evaluate the impact of coadministered influenza vaccine on the immune response to RSV-A; and to evaluate the impact of coadministered RSV vaccine on the immune response to influenza.

The main purposes of Part B of this study are to evaluate the safety, tolerability, and immunogenicity of mRNA-1345 coadministered with mRNA-1273.214; to evaluate the effect of coadministered mRNA-1273.214 on the immune response to RSV-A; and to evaluate the effect of coadministered RSV vaccine on the immune response to severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).

The main purposes of Part C (single arm, open-label) of this study are to evaluate the safety and tolerability of a booster dose (BD) of mRNA-1345 administered at 1 Year following a primary dose; to evaluate the immune response to RSV-A of a BD of mRNA 1345 administered at 1 Year following a primary dose; and to evaluate the immune response to RSV-B of a BD of mRNA-1345 administered at 1 Year following a primary dose.

ELIGIBILITY:
Key Inclusion Criteria:

Parts A and B both:

* Adults ≥50 years of age on the day of the Randomization Visit (Day 1) who are primarily responsible for self-care and activities of daily living. Participants may have one or more chronic medical diagnoses, but should be medically stable as assessed by: Absence of changes in medical therapy within 1 month due to treatment failure or toxicity; Absence of medical events qualifying as SAEs within 1 month of the planned vaccination on Day 1; and absence of known, current, and life-limiting diagnoses which, in the opinion of the investigator, would make completion of the protocol unlikely.
* Able to comply with study requirements, including access to transportation for study visits.

Part B only:

* Fully vaccinated for COVID-19 with an approved primary series according to the locally authorized or approved regimen. If the most recent COVID-19 vaccine was part of a primary series, it must be ≥ 150 days before (or less per local guidance) Day 1. If the most recent COVID-19 vaccine was a booster dose, it must be ≥ 120 days before (or less per local guidance) Day 1.

Part C:

* Participants at Part C study sites who have been enrolled in Part B (Groups 4 and 5) of this study; have immunogenicity blood sampling at Part B baseline and Day 29; completed the Day 211/end-of-study visits for Part B; were included in the per-protocol (PP) set; and received 1 dose of mRNA-1345 at least 12 months (but no later than 15 months) prior to the time of enrollment.
* Able to comply with study requirements, including access to transportation for study visits.

Key Exclusion Criteria:

Part A:

* Participant has received or plans to receive any vaccine authorized or approved by a local health agency ≤28 days prior to study injections (Day 1) or plans to receive a vaccine authorized or approved by a local health agency within 28 days after the study injections.
* Prior participation in research involving receipt of any investigational product (drug/biologic/device including any investigational RSV product) within 45 days before the planned date of the Day 1 study injection.
* Participant has received a seasonal influenza vaccine or any other investigational influenza vaccine ≤180 days prior to the Randomization Visit (Day 1).
* History of a serious reaction to any prior vaccination, or Guillain-Barré syndrome within 6 weeks of any prior influenza immunization.
* Participated in an interventional clinical study within 28 days prior to the Screening Visit based on the medical history interview or plans to do so while participating in this study.

Part B:

* Participant has received or plans to receive any vaccine authorized or approved by a local health agency ≤ 28 days prior to study injections (Day 1) or plans to receive a vaccine authorized or approved by a local health agency within 28 days after the study injections (with the exception of SARS-Cov-2 vaccination).
* Prior participation in research involving receipt of any investigational product (drug/biologic/device with the exception of RSV investigation products) within 45 days before the planned date of the Day 1 study injection.
* Prior receipt of any investigational/approved RSV product within 1 year of the Day 1 study injection.
* Has known history of SARS-CoV-2 infection within 90 days prior to enrollment.

Parts A and B both:

* Participant had significant exposure to someone with SARS-CoV-2 infection or COVID-19 in the past 10 days, as defined by the United States (US) Centers for Disease Control and Prevention (CDC) as a close contact of someone who has had COVID-19.

Part C:

* Participation in another interventional clinical research study where participant has received an investigational product (drug/biologic/device) within 6 months before the planned date of the BD Day 1 study injection. Any prior receipt of an investigational or approved vaccine against RSV, except as part of mRNA-1345 Study P302 Part B, is exclusionary.
* Participant has received or plans to receive any vaccine authorized or approved by a local health agency ≤28 days prior to the study injection (BD Day 1) or plans to receive a vaccine authorized or approved by a local health agency within 28 days after the study injections.
* History of a serious reaction to any prior vaccination or Guillain-Barré syndrome 6 weeks after any prior influenza immunization.

Other inclusion and/or exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3317 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (62):
- United States (62):
  - Central Research Associates Inc, Birmingham, Alabama
  - Del Sol Research Management - Clinedge - PPDS, Tucson, Arizona
  - Paragon Rx Clinical, Inc, Garden Grove, California
  - Ark Clinical Research, Long Beach, California
  - Long Beach Clinical Trials, LLC (Site 1), Long Beach, California
  - Long Beach Clinical Trials, LLC (Site 2), Long Beach, California
  - Central Valley Research, LLC, Modesto, California
  - Velocity Clinical Research - Panorama City, Panorama City, California
  - Empire Clinical Research, Pomona, California
  - Acclaim Clinical Research, San Diego, California
  - Medical Center For Clinical Research - M3 WR - ERN - PPDS, San Diego, California
  - Ark Clinical Research, Tustin, California
  - Chase Medical Research LLC, Waterbury, Connecticut
  - Teradan Clinical Trials, Brandon, Florida
  - Revival Research Corporation - Clinedge - PPDS, Doral, Florida
  - Dolphin Medical Research, Doral, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - Westside Center for Clinical Research - ERN - PPDS, Jacksonville, Florida
  - Suncoast Research Group LLC - ERN-PPDS, Miami, Florida
  - Suncoast Research Associates LLC - ERN - PPDS, Miami, Florida
  - Floridian Clinical Research - ClinEdge - PPDS, Miami Lakes, Florida
  - Tekton Research - Georgia - Platinum - PPDS, Chamblee, Georgia
  - Lifeline Primary Care / CCT Research, Lilburn, Georgia
  - Georgia Clinic / CCT Research, Norcross, Georgia
  - Meridian Clinical Research (Savannah Georgia) - Platinum - PPDS, Savannah, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Meridian Clinical Research (Sioux City - Iowa), Sioux City, Iowa
  - Meridian Clinical Research, LLC (Overland Park, Kansas) - Platinum - PPDS, Overland Park, Kansas
  - Meridian Clinical Research (Baton Rouge-Louisiana) - Platinum - PPDS, Baton Rouge, Louisiana
  - Clinical Trials of SWLA, LLC, Lake Charles, Louisiana
  - Meridian Clinical Research (Rockville Maryland) - Platinum - PPDS, Rockville, Maryland
  - Clinical Research Institute, Inc - CRN - PPDS, Minneapolis, Minnesota
  - Meridian Clinical Research (Grand Island) - Platinum - PPDS, Grand Island, Nebraska
  - Meridian Clinical Research, LLC (Lincoln Nebraska) - Platinum - PPDS, Lincoln, Nebraska
  - Be Well Clinical Studies, LLC, Lincoln, Nebraska
  - Meridian Clinical Research, Norfolk, Nebraska
  - Meridian Clinical Research (Omaha-Nebraska) - Platinum - PPDS, Omaha, Nebraska
  - Midwest Regional Health Services - CCT Research, Omaha, Nebraska
  - Clinical Research Center of Nevada - ERN - PPDS, Las Vegas, Nevada
  - Santa Rosa Medical Centers of Nevada - CCT Research, Las Vegas, Nevada
  - Meridian Clinical Research (Endwell-New York) - Platinum - PPDS, Endwell, New York
  - IMA Medical Research, PC., New York, New York
  - CHEAR Center LLC - ClinEdge - PPDS, The Bronx, New York
  - Javara Research Inc. - Charlotte - Javara - PPDS, Charlotte, North Carolina
  - M3 Wake Research, Inc - M3 WR - ERN - PPDS, Raleigh, North Carolina
  - Velocity Clinical Research - Cleveland - ERN - PPDS, Cleveland, Ohio
  - Meridian Clinical Research - Cincinnati - Platinum - PPDS, Springdale, Ohio
  - Tekton Research, Moore, Oklahoma
  - Velocity Clinical Research - Anderson - ERN - PPDS, Anderson, South Carolina
  - Velocity Clinical Research - Greenville - ERN - PPDS, Greenville, South Carolina
  - Trial Management Associates LLC - ERN - PPDS, Myrtle Beach, South Carolina
  - Velocity Clinical Research - Spartanburg - ERN - PPDS, Spartanburg, South Carolina
  - New Phase Research & Development, Knoxville, Tennessee
  - Benchmark Research - Austin - HyperCore - PPDS, Austin, Texas
  - Tekton Research - Beaumont - Platinum - PPDS, Beaumont, Texas
  - Zenos Clinical Research, Dallas, Texas
  - Milton Haber, M.D., Laredo, Texas
  - Sun Research Institute, San Antonio, Texas
  - Cope Family Medicine - Ogden Clinic, Bountiful, Utah
  - CCT Research at Springville Dermatology, Springville, Utah
  - Javara Inc./Privia Medical Group INC, Forest, Virginia
  - Meridian Clinical Research - Family Practice Ports - Portsmouth - Platinum - PPDS, Portsmouth, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goswami J, Cardona JF, Caso J, Hsu DC, Simorellis AK, Wilson L, Dhar R, Wang X, Kapoor A, Collins A, Righi V, Lan L, Du J, Zhou H, Stoszek SK, Shaw CA, Reuter C, Wilson E, Das R. Safety, Tolerability, and Immunogenicity of Revaccination with mRNA-1345, an mRNA Vaccine Against RSV, Administered 12 Months Following a Primary Dose in Adults Aged >/=50 Years. Clin Infect Dis. 2025 Sep 23:ciaf515. doi: 10.1093/cid/ciaf515. Online ahead of print. PMID 40988124
- [Derived] Goswami J, Cardona JF, Hsu DC, Simorellis AK, Wilson L, Dhar R, Tomassini JE, Wang X, Kapoor A, Collins A, Righi V, Lan L, Du J, Zhou H, Stoszek SK, Shaw CA, Reuter C, Wilson E, Miller JM, Das R; study investigators. Safety and immunogenicity of mRNA-1345 RSV vaccine coadministered with an influenza or COVID-19 vaccine in adults aged 50 years or older: an observer-blinded, placebo-controlled, randomised, phase 3 trial. Lancet Infect Dis. 2025 Apr;25(4):411-423. doi: 10.1016/S1473-3099(24)00589-9. Epub 2024 Nov 25. PMID 39608389

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: mRNA-1345 + Placebo: Participants received a single injection each of mRNA-1345 and placebo, administered intramuscularly (IM) on Day 1.
- Part A: mRNA-1345 + Afluria® Quadrivalent: Participants received a single injection each of mRNA-1345 and Afluria® quadrivalent, administered IM on Day 1.
- Part A: Afluria® Quadrivalent + Placebo: Participants received a single injection each of Afluria® quadrivalent and placebo, administered IM on Day 1.
- Part B: mRNA-1345 + Placebo + mRNA-1273.214: Participants received a single injection of mRNA-1345 and placebo, administered IM on Day 1.
  (Note: An additional injection of mRNA-1273.214 was administered on Day 29 to allow all study participants to receive an mRNA-1273.214 booster vaccination.)
- Part B: mRNA-1345 + mRNA-1273.214 + Placebo: Participants received a single injection each of mRNA-1345 and mRNA-1273.214, administered IM on Day 1.
  (Note: An additional injection of placebo was administered on Day 29 to maintain blinding.)
- Part B: mRNA-1273.214 + Placebo + Placebo: Participants received a single injection each of mRNA-1273.214 and placebo, administered IM on Day 1.
  (Note: An additional injection of placebo was administered on Day 29 to maintain blinding.)
- Part C: mRNA-1345 Revaccination: Participants received mRNA-1345 primary vaccination in Part B and opted to receive revaccination in Part C. Participants received a single mRNA-1345 injection at least 12 months (but not longer than 15 months) after primary vaccination.
Period: Primary
Arm/Group | Part A: mRNA-1345 + Placebo | Part A: mRNA-1345 + Afluria® Quadrivalent | Part A: Afluria® Quadrivalent + Placebo | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo | Part B: mRNA-1273.214 + Placebo + Placebo | Part C: mRNA-1345 Revaccination
Started | 249 | 690 | 692 | 560 | 564 | 562 | 0
Received at Least 1 Dose of Any Study Injection | 249 | 685 (5 randomized participants did not receive the study intervention) | 689 (3 randomized participants did not receive the study intervention) | 556 (4 randomized participants did not receive the study intervention) | 562 (2 randomized participants did not receive the study intervention) | 558 (4 randomized participants did not receive the study intervention) | 0
Part B Day 1 Injection (Part B Day 1 Injection consisted of all randomized participants who received any study injection on Day 1.) | 0 | 0 | 0 | 556 | 562 | 558 | 0
Part B Day 29 Injection (Part B Day 29 Injection consisted of all randomized participants who received any study injection on Day 29.) | 0 | 0 | 0 | 530 | 535 | 536 | 0
Safety Set (Safety Set consisted of all randomized participants who received any study intervention. Participants were included in the treatment arm corresponding to the study intervention they actually received.) | 249 | 685 | 689 | 554 | 562 | 560 | 0
Solicited Safety Set (Day 1 Injection) (Solicited Safety Set consisted of all randomized participants who received any study injection on Day 1 and contributed any solicited ARs.) | 249 | 678 | 683 | 553 | 562 | 557 | 0
Part B Solicited Safety Set Day 29 Injection (Part B Solicited Safety Set Day 29 Injection consisted of all randomized participants who received any study injection on Day 29 and contributed any solicited ARs.) | 0 | 0 | 0 | 522 | 532 | 528 | 0
Per-protocol (PP) Set (PP Set consisted of all participants who received the assigned study injections according to protocol, complied with immunogenicity sampling, and had no major protocol deviations.) | 232 | 639 | 626 | 513 | 514 | 519 | 0
Completed | 233 | 652 | 643 | 500 | 516 | 510 | 0
Not Completed | 16 | 38 | 49 | 60 | 48 | 52 | 0
Not completed — Lost to Follow-up | 12 | 21 | 38 | 30 | 25 | 28 | 0
Not completed — Withdrawal by Subject | 4 | 11 | 8 | 23 | 20 | 19 | 0
Not completed — Protocol Violation | 0 | 2 | 0 | 4 | 0 | 3 | 0
Not completed — Death | 0 | 3 | 1 | 1 | 0 | 0 | 0
Not completed — Other Than Specified | 0 | 1 | 2 | 1 | 2 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Revaccination
Arm/Group | Part A: mRNA-1345 + Placebo | Part A: mRNA-1345 + Afluria® Quadrivalent | Part A: Afluria® Quadrivalent + Placebo | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo | Part B: mRNA-1273.214 + Placebo + Placebo | Part C: mRNA-1345 Revaccination
Started | 0 | 0 | 0 | 0 | 0 | 0 | 543
Part C Safety Set (Part C Safety Set consisted of all enrolled participants who received any revaccination of mRNA-1345.) | 0 | 0 | 0 | 0 | 0 | 0 | 543
Part C Solicited Safety Set (Part C Solicited Safety Set consisted of all enrolled participants who received revaccination of mRNA-1345 and contributed any solicited ARs.) | 0 | 0 | 0 | 0 | 0 | 0 | 543
Part C PP Set (Part C PP Set consisted of all enrolled participants who received planned revaccination of mRNA-1345, had prevaccination and at least 1 revaccination Day 29 assessment of immunogenicity, complied with immunogenicity sampling, and had no major protocol deviations.) | 0 | 0 | 0 | 0 | 0 | 0 | 525
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 525
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 18
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Randomized Set included all participants who were randomized in the study, regardless of the participant's treatment status in the study.
Groups:
- Part A: mRNA-1345 + Placebo: Participants received a single injection each of mRNA-1345 and placebo, administered IM on Day 1.
- Total: Total of all reporting groups
Arm/Group | Part A: mRNA-1345 + Placebo | Part A: mRNA-1345 + Afluria® Quadrivalent | Part A: Afluria® Quadrivalent + Placebo | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo | Part B: mRNA-1273.214 + Placebo + Placebo | Total
Number analyzed (Participants) | 249 | 690 | 692 | 560 | 564 | 562 | 3317
Age, Customized [Number; unit: years]
  ≥50 years of age | 249 | 690 | 692 | 560 | 564 | 562 | 3317
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 367 | 375 | 315 | 317 | 296 | 1811
  Male | 108 | 323 | 317 | 245 | 247 | 266 | 1506
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 91 | 240 | 249 | 213 | 214 | 223 | 1230
  Not Hispanic or Latino | 158 | 445 | 442 | 342 | 349 | 333 | 2069
  Unknown or Not Reported | 0 | 5 | 1 | 5 | 1 | 6 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 189 | 524 | 514 | 430 | 428 | 438 | 2523
  Race: Black or African American | 59 | 157 | 166 | 112 | 113 | 111 | 718
  Race: Asian | 0 | 4 | 3 | 6 | 8 | 1 | 22
  Race: American Indian or Alaska Native | 1 | 1 | 4 | 6 | 4 | 2 | 18
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 3 | 1 | 3 | 0 | 8
  Race: Other | 0 | 1 | 1 | 1 | 0 | 3 | 6
  Race: Multiple | 0 | 2 | 0 | 1 | 0 | 3 | 6
  Race: Not Reported | 0 | 0 | 1 | 3 | 8 | 4 | 16

OUTCOME MEASURES:

1. Secondary Outcome: Part A: GMT of Serum RSV-B NAbs at Day 29
Description: Antibody values reported as below LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ were replaced by the ULOQ. LLOQ was 10 IU/mL and ULOQ was 112476 for RSV-B. As prespecified, only arms where participants received mRNA-1345 are presented for this outcome measure.
Time Frame: Day 29
Population: PP Set: All participants who received the assigned study injections according to protocol, complied with immunogenicity sampling (baseline and at least 1 Day 29 post-injection assessment), and have no major protocol deviations affecting the immune response. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Part A: mRNA-1345 + Placebo | Part A: mRNA-1345 + Afluria® Quadrivalent
Number analyzed (Participants) | 232 | 639
IU/mL | 10436.03 [8973.29 to 12137.20] | 8909.80 [8016.02 to 9903.24]
Statistical Analysis 1: Comparison: Part A: mRNA-1345 + Placebo vs Part A: mRNA-1345 + Afluria® Quadrivalent; Test type: Non-Inferiority — Lower bound of the 95% CI of GMR >0.667, using a noninferiority margin of 1.5; GMR = 0.854, 95% CI 2-sided [0.728 to 1.002] — mRNA-1345+Afluria group compared mRNA-1345 alone group

2. Secondary Outcome: Part A: Percentage of Participants With Seroresponse in RSV-B NAbs at Day 29
Description: Seroresponse was defined as ≥4 × LLOQ if baseline was <LLOQ or 4-fold or greater increase from baseline if baseline was ≥LLOQ. As prespecified, only arms where participants received mRNA-1345 are presented for this outcome measure.
Time Frame: Day 29
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: mRNA-1345 + Placebo | Part A: mRNA-1345 + Afluria® Quadrivalent
Number analyzed (Participants) | 232 | 639
percentage of participants | 63.8 [57.2 to 70.0] | 49.5 [45.5 to 53.4]
Statistical Analysis 1: Comparison: Part A: mRNA-1345 + Placebo vs Part A: mRNA-1345 + Afluria® Quadrivalent; Test type: Non-Inferiority — Lower bound of the 95% CI of the SRR difference >-10%, using noninferiority margin of 10%; Difference = -14.3, 95% CI 2-sided [-21.5 to -6.9] — mRNA-1345+Afluria group compared mRNA-1345 alone group

3. Secondary Outcome: Part A: Percentage of Participants With Seroconversion in Influenza A and B Strains at Day 181
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Washington and Phuket strains. Seroconversion was defined as a titer ≥1:40 if baseline was <1:10 or a 4-fold or greater rise from baseline in the titers if Baseline was ≥1:10. As prespecified, only arms where participants received Afluria® Quadrivalent are presented for this outcome measure.
Time Frame: Day 181
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: mRNA-1345 + Afluria® Quadrivalent | Part A: Afluria® Quadrivalent + Placebo
Number analyzed (Participants) | 609 | 595
percentage of participants
  Influenza A H1N1 Antibody | 41.1 [37.1 to 45.1] | 38.8 [34.9 to 42.9]
  Influenza A H3N2 Antibody | 29.4 [25.8 to 33.2] | 28.7 [25.1 to 32.6]
  Influenza B Washington Antibody | 19.5 [16.5 to 22.9] | 19.7 [16.5 to 23.1]
  Influenza B Phuket Antibody | 17.2 [14.3 to 20.5] | 18.8 [15.8 to 22.2]

4. Secondary Outcome: Part A: GMT of Serum RSV-A and RSV-B NAbs at Day 181
Description: Antibody values reported as below LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ were replaced by the ULOQ. LLOQ was 13 IU/mL and ULOQ was 259061 IU/mL for RSV-A. LLOQ was 10 IU/mL and ULOQ was 112476 for RSV-B. As prespecified, only arms where participants received mRNA-1345 are presented for this outcome measure.
Time Frame: Day 181
Population: PP Set: All participants who received the assigned study injections according to protocol, complied with immunogenicity sampling (baseline and at least 1 Day 29 post-injection assessment), and have no major protocol deviations affecting the immune response. 'Overall number of participants analyzed' = participants evaluable for this endpoint. Number analyzed' = participants evaluable for specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Part A: mRNA-1345 + Placebo | Part A: mRNA-1345 + Afluria® Quadrivalent
Number analyzed (Participants) | 218 | 613
IU/mL
  RSV-A: number analyzed (Participants) | 218 | 612
  RSV-A | 7551.13 [6504.13 to 8766.68] | 6429.48 [5850.16 to 7066.17]
  RSV-B | 2402.86 [2120.18 to 2723.23] | 2301.47 [2114.95 to 2504.44]

5. Secondary Outcome: Part A: Geometric Mean Fold Rise (GMFR) of Serum RSV-A and RSV-B NAbs at Day 181
Description: 95% CI for GMFR (postinjection/baseline titers) was calculated based on the t-distribution of the differences in the log-transformed values between analysis timepoint and baseline, then back transformed to the original scale for presentation. As prespecified, only arms where participants received mRNA-1345 are presented for this outcome measure.
Time Frame: Day 181
Population: PP Set: All participants who received the assigned study injections according to protocol, complied with immunogenicity sampling (baseline and at least 1 Day 29 post-injection assessment), and had no major protocol deviations affecting the immune response. 'Overall number of participants analyzed' = participants evaluable for this endpoint. 'Number analyzed' = participants evaluable for specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part A: mRNA-1345 + Placebo | Part A: mRNA-1345 + Afluria® Quadrivalent
Number analyzed (Participants) | 218 | 613
ratio
  RSV-A: number analyzed (Participants) | 218 | 612
  RSV-A | 3.46 [2.97 to 4.04] | 2.19 [1.99 to 2.40]
  RSV-B | 1.32 [1.17 to 1.49] | 0.94 [0.87 to 1.02]

6. Secondary Outcome: Part A: Percentage of Participants With Seroresponse in RSV-A and RSV-B NAb Titers at Day 181
Description: Seroresponse was defined as ≥4 × LLOQ if baseline was <LLOQ or 4-fold or greater increase from baseline if baseline was ≥LLOQ.As prespecified, only arms where participants received mRNA-1345 are presented for this outcome measure.
Time Frame: Day 181
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: mRNA-1345 + Placebo | Part A: mRNA-1345 + Afluria® Quadrivalent
Number analyzed (Participants) | 218 | 613
percentage of participants
  RSV-A: number analyzed (Participants) | 218 | 612
  RSV-A | 46.8 [40.0 to 53.6] | 29.9 [26.3 to 33.7]
  RSV-B | 13.3 [9.1 to 18.5] | 6.7 [4.8 to 9.0]

7. Secondary Outcome: Part A: Percentage of Participants With ≥2-fold Increases From Baseline in RSV-A and RSV-B NAb Titers at Day 181
Description: ≥2-fold increase from baseline at participant level was defined as a change from below the LLOQ to equal or above 2 * LLOQ, or at least a 2-fold increase if baseline was equal to or above the LLOQ. As prespecified, only arms where participants received mRNA-1345 are presented for this outcome measure.
Time Frame: Baseline to Day 181
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: mRNA-1345 + Placebo | Part A: mRNA-1345 + Afluria® Quadrivalent
Number analyzed (Participants) | 218 | 613
percentage of participants
  RSV-A: number analyzed (Participants) | 218 | 612
  RSV-A | 67.0 [60.3 to 73.2] | 54.1 [50.0 to 58.1]
  RSV-B | 32.1 [26.0 to 38.7] | 21.0 [17.9 to 24.5]

8. Secondary Outcome: Part A: GMT of Serum Anti-HA Ab Level, as Measured by HAI Assay for Influenza at Day 181
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Washington and Phuket strains. Antibody values reported as below LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ were replaced by the ULOQ. LLOQ was 10 and ULOQ was 2560 for Influenza A. LLOQ was 10 and ULOQ was 640 for Influenza B. As prespecified, only arms where participants received Afluria® Quadrivalent are presented for this outcome measure.
Time Frame: Day 181
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A: mRNA-1345 + Afluria® Quadrivalent | Part A: Afluria® Quadrivalent + Placebo
Number analyzed (Participants) | 613 | 601
titer
  Influenza A H1N1 Antibody | 155.59 [138.10 to 175.31] | 156.47 [139.65 to 175.33]
  Influenza A H3N2 Antibody | 113.58 [101.54 to 127.06] | 109.36 [98.28 to 121.68]
  Influenza B Washington Antibody | 32.11 [29.10 to 35.43] | 35.03 [31.76 to 38.64]
  Influenza B Phuket Antibody | 25.64 [23.34 to 28.17] | 26.43 [24.17 to 28.91]

9. Secondary Outcome: Part A: GMFR of Serum Anti-HA Ab Level, as Measured by HAI Assay for Influenza at Day 181
Description: Influenza A strains included H1N1 and H3N2 and influenza B strains included Washington and Phuket strains. Antibody values reported as below LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ were replaced by the ULOQ. LLOQ was 10 and ULOQ was 2560 for Influenza A. LLOQ was 10 and ULOQ was 640 for Influenza B. 95% CI for GMFR (postinjection/baseline titers) was calculated based on the t-distribution of the differences in the log-transformed values between analysis timepoint and baseline, then back transformed to the original scale for presentation. As prespecified, only arms where participants received Afluria® Quadrivalent are presented for this outcome measure.
Time Frame: Day 181
Population: PP Set: All participants who received the assigned study injections according to protocol, complied with immunogenicity sampling (baseline and at least 1 Day 29 post-injection assessment), and had no major protocol deviations affecting the immune response. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part A: mRNA-1345 + Afluria® Quadrivalent | Part A: Afluria® Quadrivalent + Placebo
Number analyzed (Participants) | 609 | 595
ratio
  Influenza A H1N1 Antibody | 3.21 [2.80 to 3.68] | 3.08 [2.70 to 3.51]
  Influenza A H3N2 Antibody | 2.28 [2.04 to 2.55] | 2.23 [2.00 to 2.49]
  Influenza B Washington Antibody | 1.80 [1.66 to 1.96] | 1.95 [1.79 to 2.13]
  Influenza B Phuket Antibody | 1.76 [1.63 to 1.90] | 1.79 [1.66 to 1.93]

10. Secondary Outcome: Part B: GMT of Serum RSV-B NAbs at Day 29
Description: as for outcome 1
Time Frame: Day 29
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo
Number analyzed (Participants) | 511 | 513
IU/mL | 6584.54 [5961.73 to 7272.40] | 5843.94 [5292.14 to 6453.28]
Statistical Analysis 1: Comparison: Part B: mRNA-1345 + Placebo + mRNA-1273.214 vs Part B: mRNA-1345 + mRNA-1273.214 + Placebo; Test type: Non-Inferiority — Lower bound of the 95% CI of GMR >0.667, using a noninferiority margin of 1.5; GMR = 0.888, 95% CI 2-sided [0.791 to 0.995] — mRNA-1345+mRNA-1273.214 compared with mRNA-1345 alone

11. Secondary Outcome: Part B: Percentage of Participants With Seroresponse in RSV-B NAbs From Baseline to Day 29
Description: as for outcome 2
Time Frame: Baseline to Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo
Number analyzed (Participants) | 511 | 513
percentage of participants | 51.9 [47.4 to 56.3] | 46.0 [41.6 to 50.4]
Statistical Analysis 1: Comparison: Part B: mRNA-1345 + Placebo + mRNA-1273.214 vs Part B: mRNA-1345 + mRNA-1273.214 + Placebo; Test type: Non-Inferiority — Lower bound of the 95% CI of the SRR difference >-10%, using noninferiority margin of 10%; Difference = -5.9, 95% CI 2-sided [-11.9 to 0.3] — mRNA-1345+mRNA-1273.214 compared with mRNA-1345 alone

12. Secondary Outcome: Part B: GMT of Serum RSV-A and RSV-B NAbs at Day 181
Description: as for outcome 4
Time Frame: Day 181
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo
Number analyzed (Participants) | 476 | 487
IU/mL
  RSV-A | 6456.32 [5830.84 to 7148.91] | 5221.87 [4723.14 to 5773.26]
  RSV-B | 2447.67 [2236.91 to 2678.28] | 2274.83 [2070.95 to 2498.79]

13. Secondary Outcome: Part B: GMFR of Serum RSV-A and RSV-B NAbs at Day 181
Description: Antibody values reported as below LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ were replaced by the ULOQ. As prespecified, only arms where participants received mRNA-1345 are presented for this outcome measure.
Time Frame: Day 181
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo
Number analyzed (Participants) | 476 | 487
ratio
  RSV-A | 2.91 [2.65 to 3.20] | 2.58 [2.36 to 2.82]
  RSV-B: number analyzed (Participants) | 475 | 487
  RSV-B | 1.61 [1.48 to 1.75] | 1.49 [1.38 to 1.61]

14. Secondary Outcome: Part B: GMC of Serum Ab Level, as Measured by Neutralization Assay for SARS-Cov-2 at Day 181
Description: 95% CI for GM value was calculated based on the t-distribution of the log-transformed values between analysis timepoint and baseline, then back transformed to the original scale for presentation. SARS-CoV-2 variants included Wuhan-Hu-1 and B.1.1.529. Antibody values reported as below LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ were replaced by the ULOQ. LLOQ was 10 AU/mL and ULOQ was 111433 AU/mL for Wuhan-Hu-1. LLOQ was 8 AU/mL and ULOQ was 24503 for B1.1.529.
Time Frame: Day 181
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo | Part B: mRNA-1273.214 + Placebo + Placebo
Number analyzed (Participants) | 476 | 485 | 486
AU/mL
  Wuhan-Hu-1 | 4075.34 [3722.53 to 4461.58] | 3615.45 [3272.04 to 3994.91] | 3665.39 [3335.37 to 4028.07]
  B.1.1.529 | 1002.35 [894.17 to 1123.61] | 889.75 [791.84 to 999.76] | 919.49 [820.46 to 1030.46]

15. Secondary Outcome: Part B: GMFR of Serum Ab Level, as Measured by Neutralization Assay for SARS-Cov-2 at Day 181
Description: 95% CI for GMFR (postinjection/baseline titers) was calculated based on the t-distribution of the differences in the log-transformed values between analysis timepoint and baseline, then back transformed to the original scale for presentation.
Time Frame: Day 181
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo | Part B: mRNA-1273.214 + Placebo + Placebo
Number analyzed (Participants) | 476 | 485 | 486
ratio
  Wuhan-Hu-1: number analyzed (Participants) | 474 | 479 | 484
  Wuhan-Hu-1 | 2.12 [1.90 to 2.38] | 1.94 [1.72 to 2.19] | 1.84 [1.65 to 2.06]
  B.1.1.529 | 3.57 [3.12 to 4.09] | 3.27 [2.83 to 3.78] | 3.13 [2.75 to 3.55]

16. Secondary Outcome: Part B: Percentage of Participants With Seroresponse for SARS-Cov-2 NAbs From Baseline to Day 181
Description: Seroresponse was defined as ≥4 × LLOQ if baseline was <LLOQ or 4-fold or greater increase from baseline if baseline was ≥LLOQ. SARS-CoV-2 variants included Wuhan-Hu-1 and B.1.1.529. Antibody values reported as below LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ were replaced by the ULOQ. LLOQ was 10 and ULOQ was 111433 for Wuhan-Hu-1. LLOQ was 8 and ULOQ was B.1.1.529 for B1.1.529.
Time Frame: Baseline to Day 181
Population: PP Set: All participants who received the assigned study injections according to protocol, complied with immunogenicity sampling (baseline and at least 1 Day 29 post-injection assessment), and had no major protocol deviations affecting the immune response. 'Overall number of participants analyzed' = participants evaluable for this endpoint. Number analyzed' = participants evaluable for specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo | Part B: mRNA-1273.214 + Placebo + Placebo
Number analyzed (Participants) | 476 | 485 | 486
percentage of participants
  Wuhan-Hu-1: number analyzed (Participants) | 474 | 479 | 484
  Wuhan-Hu-1 | 24.1 [20.3 to 28.2] | 23.6 [19.9 to 27.7] | 19.8 [16.4 to 23.7]
  B.1.1.529 | 44.7 [40.2 to 49.3] | 41.0 [36.6 to 45.6] | 40.5 [36.1 to 45.0]

17. Secondary Outcome: Part B: Percentage of Participants With Seroresponse in RSV-A and RSV-B NAb Titers at Day 181
Description: as for outcome 2
Time Frame: Day 181
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo
Number analyzed (Participants) | 476 | 487
percentage of participants
  RSV-A: number analyzed (Participants) | 476 | 486
  RSV-A | 34.9 [30.6 to 39.3] | 30.2 [26.1 to 34.5]
  RSV-B: number analyzed (Participants) | 475 | 487
  RSV-B | 14.9 [11.9 to 18.5] | 12.7 [9.9 to 16.0]

18. Secondary Outcome: Part B: Percentage of Participants With ≥2-fold Increases From Baseline in RSV-A and RSV-B NAb Titers at Day 181
Description: ≥2-fold increase from baseline at participant level was defined as a change from below the LLOQ to equal or above 2 * LLOQ, or at least a 2-fold increase if baseline was equal to or above the LLOQ. LLOQ was 13 IU/mL and ULOQ was 259061 IU/mL for RSV-A. LLOQ was 10 IU/mL and ULOQ was 112476 for RSV-B. As prespecified, only arms where participants received mRNA-1345 are presented for this outcome measure.
Time Frame: Baseline to Day 181
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo
Number analyzed (Participants) | 476 | 487
percentage of participants
  RSV-A | 62.8 [58.3 to 67.2] | 58.3 [53.8 to 62.7]
  RSV-B: number analyzed (Participants) | 475 | 487
  RSV-B | 36.4 [32.1 to 40.9] | 35.7 [31.5 to 40.2]

19. Secondary Outcome: Part B: GMT of Serum RSV-A and RSV-B NAbs at Day 211
Description: as for outcome 4
Time Frame: Day 211
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo
Number analyzed (Participants) | 474 | 487
IU/mL
  RSV-A | 5921.09 [5357.33 to 6544.17] | 4696.74 [4245.92 to 5195.44]
  RSV-B: number analyzed (Participants) | 473 | 487
  RSV-B | 2261.26 [2069.70 to 2470.56] | 2132.70 [1943.36 to 2340.49]

20. Secondary Outcome: Part B: GMFR of Serum RSV-A and RSV-B NAbs at Day 211
Description: as for outcome 13
Time Frame: Day 211
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo
Number analyzed (Participants) | 474 | 487
ratio
  RSV-A: number analyzed (Participants) | 474 | 486
  RSV-A | 2.71 [2.48 to 2.98] | 2.35 [2.15 to 2.56]
  RSV-B: number analyzed (Participants) | 472 | 487
  RSV-B | 1.50 [1.39 to 1.63] | 1.40 [1.30 to 1.51]

21. Secondary Outcome: Part B: GMC of Serum Ab Level, as Measured by Neutralization Assay for SARS-Cov-2 at Day 211
Description: as for outcome 14
Time Frame: Day 211
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo | Part B: mRNA-1273.214 + Placebo + Placebo
Number analyzed (Participants) | 471 | 485 | 486
AU/mL
  Wuhan-Hu-1 | 3551.74 [3245.10 to 3887.35] | 3034.11 [2743.48 to 3355.54] | 3123.69 [2841.55 to 3433.84]
  B.1.1.529 | 923.10 [826.89 to 1030.51] | 797.17 [708.18 to 897.33] | 795.90 [709.19 to 893.21]

22. Secondary Outcome: Part B: GMFR of Serum Ab Level, as Measured by Neutralization Assay for SARS-Cov-2 at Day 211
Description: as for outcome 15
Time Frame: Day 211
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo | Part B: mRNA-1273.214 + Placebo + Placebo
Number analyzed (Participants) | 471 | 485 | 486
ratio
  Wuhan-Hu-1: number analyzed (Participants) | 469 | 479 | 484
  Wuhan-Hu-1 | 1.87 [1.66 to 2.09] | 1.64 [1.45 to 1.85] | 1.59 [1.42 to 1.77]
  B.1.1.529 | 3.31 [2.90 to 3.79] | 2.95 [2.56 to 3.40] | 2.72 [2.39 to 3.10]

23. Secondary Outcome: Part B: Percentage of Participants With Seroresponse for SARS-Cov-2 NAbs at Day 211
Description: as for outcome 16
Time Frame: Day 211
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo | Part B: mRNA-1273.214 + Placebo + Placebo
Number analyzed (Participants) | 471 | 485 | 486
percentage of participants
  Wuhan-Hu-1: number analyzed (Participants) | 469 | 479 | 484
  Wuhan-Hu-1 | 21.1 [17.5 to 25.1] | 20.3 [16.7 to 24.1] | 17.8 [14.5 to 21.5]
  B.1.1.529 | 41.4 [36.9 to 46.0] | 38.8 [34.4 to 43.3] | 37.0 [32.7 to 41.5]

24. Secondary Outcome: Part B: Percentage of Participants With Seroresponse in RSV-A and RSV-B NAb Titers at Day 211
Description: as for outcome 2
Time Frame: Day 211
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo
Number analyzed (Participants) | 474 | 487
percentage of participants
  RSV-A: number analyzed (Participants) | 474 | 486
  RSV-A | 32.5 [28.3 to 36.9] | 26.5 [22.7 to 30.7]
  RSV-B: number analyzed (Participants) | 472 | 487
  RSV-B | 12.3 [9.5 to 15.6] | 10.1 [7.5 to 13.1]

25. Secondary Outcome: Part B: Percentage of Participants With ≥2-fold Increases From Baseline in RSV-A and RSV-B NAb Titers at Day 211
Description: as for outcome 18
Time Frame: Day 211
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo
Number analyzed (Participants) | 474 | 487
percentage of participants
  RSV-A: number analyzed (Participants) | 474 | 486
  RSV-A | 57.8 [53.2 to 62.3] | 53.7 [49.2 to 58.2]
  RSV-B: number analyzed (Participants) | 472 | 487
  RSV-B | 33.7 [29.4 to 38.1] | 30.6 [26.5 to 34.9]

26. Secondary Outcome: Part C: Percentage of Participants With Seroresponse in RSV-A and RSV-B NAbs From Baseline (Before Primary Vaccination) to Revaccination Day 29
Description: Seroresponse was defined as ≥4 × LLOQ if baseline was <LLOQ or 4-fold or greater increase from baseline if baseline was ≥LLOQ. Primary vaccination Day 29 (received in Part B) and Revaccination Day 29 are presented.
Time Frame: Baseline (Before Primary Vaccination in Part B) to Revaccination Day 29
Population: PP Set: All participants received mRNA-1345 revaccination, had prerevaccination and at least 1 postinjection assessment of immunogenicity after revaccination, complied with immunogenicity testing schedule, and had no major protocol derivations. 'Overall number of participants analyzed' = participants evaluable for this endpoint. 'Number analyzed' = participants evaluable for specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part C: mRNA-1345 Primary Vaccination: Overall participants who received a single mRNA-1345 primary vaccination in Part B and enrolled in Part C.
- Part C: mRNA-1345 Revaccincation: Participants received a single mRNA-1345 primary vaccination on Day 1 in Part B and then received revaccination with a single mRNA-1345 injection at least 12 months later (but not longer than 15 months) (Revaccination Day 1).
Arm/Group | Part C: mRNA-1345 Primary Vaccination | Part C: mRNA-1345 Revaccincation
Number analyzed (Participants) | 523 | 524
percentage of participants
  RSV-A: number analyzed (Participants) | 518 | 524
  RSV-A | 75.3 [71.3 to 78.9] | 77.5 [73.7 to 81.0]
  RSV-B | 48.2 [43.8 to 52.6] | 47.5 [43.2 to 51.9]

27. Secondary Outcome: Part C: GMT of Serum RSV-A and RSV-B NAbs at Revaccination Day 361
Description: Antibody values reported as below LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ were replaced by the ULOQ. LLOQ was 13 IU/mL and ULOQ was 259061 IU/mL for RSV-A. LLOQ was 10 IU/mL and ULOQ was 112476 IU/mL for RSV-B.
Time Frame: Revaccination Day 361
Population: PP Set: All participants who received mRNA-1345 revaccination, had prerevaccination and at least 1 postinjection assessment of immunogenicity after revaccination, complied with immunogenicity testing schedule, and had no major protocol derivations. 'Overall number of participants analyzed' = participants evaluable for this endpoint. 'Number analyzed' = participants evaluable for specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Part C: mRNA-1345 Revaccincation
Number analyzed (Participants) | 497
IU/mL
  RSV-A: number analyzed (Participants) | 493
  RSV-A | 4708.27 [4279.78 to 5179.67]
  RSV-B | 2251.24 [2054.09 to 2467.32]

28. Secondary Outcome: Part C: GMFR of Serum RSV-A and RSV-B NAbs at Revaccination Day 361
Description: as for outcome 15
Time Frame: Revaccination Day 361
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part C: mRNA-1345 Revaccincation
Number analyzed (Participants) | 496
ratio
  RSV-A: number analyzed (Participants) | 492
  RSV-A | 2.26 [2.06 to 2.48]
  RSV-B | 1.42 [1.31 to 1.53]

29. Secondary Outcome: Part C: Percentage of Participants With Seroresponse in RSV-A and RSV-B NAbs at Revaccination Day 361
Description: Seroresponse was defined as ≥4 × LLOQ if baseline was <LLOQ or 4-fold or greater increase from baseline if baseline was ≥LLOQ.
Time Frame: Baseline to Revaccination Day 361
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part C: mRNA-1345 Revaccincation
Number analyzed (Participants) | 496
percentage of participants
  RSV-A: number analyzed (Participants) | 492
  RSV-A | 25.8 [22.0 to 29.9]
  RSV-B | 11.5 [8.8 to 14.6]

30. Secondary Outcome: Part C: Percentage of Participants With ≥2-fold Increases From Baseline (Before Primary Vaccination) in RSV-A and RSV-B NAb Titers at Revaccination Day 361
Description: ≥2-fold increase from baseline at participant level was defined as a change from below the LLOQ to equal or above 2 * LLOQ, or at least a 2-fold increase if baseline was equal to or above the LLOQ. LLOQ was 13 IU/mL and ULOQ was 259061 IU/mL for RSV-A. LLOQ was 10 IU/mL and ULOQ was 112476 IU/mL for RSV-B.
Time Frame: Baseline to Revaccination Day 361
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part C: mRNA-1345 Revaccincation
Number analyzed (Participants) | 496
percentage of participants
  RSV-A: number analyzed (Participants) | 492
  RSV-A | 53.0 [48.5 to 57.5]
  RSV-B | 32.7 [28.5 to 37.0]

31. Primary Outcome: Part A: Number of Participants With Solicited Local and Systemic Adverse Reactions (ARs) Within 7 Days After Day 1 Injection
Description: Solicited ARs were collected in an electronic diary (eDiary). Local ARs: injection site pain, erythema (redness), swelling/induration (hardness); and axillary (underarm) swelling or tenderness ipsilateral to the side of injection. Systemic ARs: fever, headache, fatigue, myalgia, arthralgia, nausea/vomiting, and chills. Note, not all solicited ARs were considered adverse events (AEs). Investigator reviewed whether the solicited AR was also to be recorded as an AE. A Summary of serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Within 7 days after Day 1 injection
Population: Solicited Safety Set included all randomized participants who received any study intervention and contributed any solicited ARs data from the time of study injection on Day 1 through the following 6 days. Participants were included in the treatment arm corresponding to the study drug they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: mRNA-1345 + Placebo | Part A: mRNA-1345 + Afluria® Quadrivalent | Part A: Afluria® Quadrivalent + Placebo
Number analyzed (Participants) | 249 | 678 | 683
Participants | 147 | 395 | 291

32. Primary Outcome: Part A: Number of Participants With Unsolicited Adverse Events (AEs) After Day 1 Injection
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Any abnormal laboratory test result (hematology, clinical chemistry, or prothrombin time [PT]/partial thromboplastin time [PTT]) or other safety assessment (for example, electrocardiogram, radiological scan, vital sign measurement), including one that worsened from baseline and was considered clinically significant in the medical and scientific judgment of the Investigator was recorded as an AE. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Day 1 through Day 28 (28 days after Day 1 injection)
Population: The Safety Set included all randomized participants who received any study intervention. Participants were included in the treatment arm corresponding to the study drug they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: mRNA-1345 + Placebo | Part A: mRNA-1345 + Afluria® Quadrivalent | Part A: Afluria® Quadrivalent + Placebo
Number analyzed (Participants) | 249 | 685 | 689
Participants | 21 | 57 | 46

33. Primary Outcome: Part A: Number of Participants With Medically Attended AEs (MAAEs), SAEs, Adverse Events of Special Interest (AESIs), and AEs Leading to Withdrawal
Description: A MAAE is an AE that leads to an unscheduled visit to a healthcare practitioner. An AESI is an AE (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor are required. An SAE was defined as any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability, was a congenital anomaly/birth defect, or was an important medical event. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Day 1 through Day 181 (end of Study Part A)
Population: as for outcome 32
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: mRNA-1345 + Placebo | Part A: mRNA-1345 + Afluria® Quadrivalent | Part A: Afluria® Quadrivalent + Placebo
Number analyzed (Participants) | 249 | 685 | 689
Participants
  MAAE | 41 | 136 | 114
  SAE | 4 | 28 | 24
  AESI | 0 | 1 | 1
  AEs Leading to Withdrawal | 0 | 3 | 1

34. Primary Outcome: Part A: Geometric Mean Titer (GMT) of Serum Respiratory Syncytial Virus Subtype A (RSV-A) Neutralizing Antibodies (NAbs) at Day 29
Description: Antibody values reported as below lower limit of quantification (LLOQ) were replaced by 0.5*LLOQ. Values greater than the upper limit of quantification (ULOQ) were replaced by the ULOQ. LLOQ was 13 international units (IU)/milliliter (mL) and ULOQ was 259061 IU/mL for RSV-A. As prespecified, only arms where participants received mRNA-1345 are presented for this outcome measure.
Time Frame: Day 29
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Part A: mRNA-1345 + Placebo | Part A: mRNA-1345 + Afluria® Quadrivalent
Number analyzed (Participants) | 232 | 639
IU/mL | 17271.72 [14448.78 to 20646.20] | 13929.98 [12291.04 to 15787.47]
Statistical Analysis 1: Comparison: Part A: mRNA-1345 + Placebo vs Part A: mRNA-1345 + Afluria® Quadrivalent; Test type: Non-Inferiority — Lower bound of the 95% CI of geometric mean ratio (GMR) >0.667, using a noninferiority margin of 1.5; GMR = 0.807, 95% CI 2-sided [0.668 to 0.974] — mRNA-1345+Afluria group compared mRNA-1345 alone group

35. Primary Outcome: Part A: Percentage of Participants With Seroresponse in RSV-A NAbs at Day 29
Description: Seroresponse was defined as ≥4 × lower limit of quantification (LLOQ) if baseline was <LLOQ or 4-fold or greater increase from baseline if baseline was ≥LLOQ. As prespecified, only arms where participants received mRNA-1345 are presented for this outcome measure.
Time Frame: Day 29
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: mRNA-1345 + Placebo | Part A: mRNA-1345 + Afluria® Quadrivalent
Number analyzed (Participants) | 232 | 639
percentage of participants | 72.4 [66.2 to 78.1] | 61.2 [57.3 to 65.0]
Statistical Analysis 1: Comparison: Part A: mRNA-1345 + Placebo vs Part A: mRNA-1345 + Afluria® Quadrivalent; Test type: Non-Inferiority — Lower bound of the 95% CI of the SRR difference >-10%, using noninferiority margin of 10%; Difference = -11.2, 95% CI 2-sided [-17.9 to -4.1] — mRNA-1345+Afluria group compared mRNA-1345 alone group

36. Primary Outcome: Part A: GMT of Serum Anti-hemagglutination (HA) Ab Level, as Measured by Hemagglutination Inhibition (HAI) Assay for Influenza at Day 29
Description: as for outcome 8
Time Frame: Day 29
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A: mRNA-1345 + Afluria® Quadrivalent | Part A: Afluria® Quadrivalent + Placebo
Number analyzed (Participants) | 630 | 619
titer
  Influenza A H1N1 Antibody | 271.27 [239.71 to 306.99] | 303.92 [268.24 to 344.35]
  Influenza A H3N2 Antibody | 144.14 [130.37 to 159.36] | 148.69 [134.35 to 164.55]
  Influenza B Washington Antibody | 57.59 [52.01 to 63.77] | 62.13 [56.05 to 68.86]
  Influenza B Phuket Antibody | 38.52 [34.91 to 42.50] | 42.40 [38.39 to 46.82]
Statistical Analysis 1: Comparison: Part A: mRNA-1345 + Afluria® Quadrivalent vs Part A: Afluria® Quadrivalent + Placebo; Influenza A H1N1 Antibody; Test type: Non-Inferiority — Lower bound of the 95% CI of GMR >0.667, using a noninferiority margin of 1.5; GMR = 0.893, 95% CI 2-sided [0.772 to 1.032] — mRNA-1345+Afluria group at Day 29 compared with the GMT of anti-HA Ab in the Afluria alone group
Statistical Analysis 2: Comparison: Part A: mRNA-1345 + Afluria® Quadrivalent vs Part A: Afluria® Quadrivalent + Placebo; Influenza A H3N2 Antibody; Test type: Non-Inferiority — Lower bound of the 95% CI of geometric mean ratio (GMR) >0.667, using a noninferiority margin of 1.5; GMR = 0.969, 95% CI 2-sided [0.861 to 1.091] — mRNA-1345+Afluria group at Day 29 compared with the GMT of anti-HA Ab in the Afluria alone group
Statistical Analysis 3: Comparison: Part A: mRNA-1345 + Afluria® Quadrivalent vs Part A: Afluria® Quadrivalent + Placebo; Influenza B Washington Antibody; Test type: Non-Inferiority — Lower bound of the 95% CI of geometric mean ratio (GMR) >0.667, using a noninferiority margin of 1.5; GMR = 0.927, 95% CI 2-sided [0.822 to 1.045] — mRNA-1345+Afluria group at Day 29 compared with the GMT of anti-HA Ab in the Afluria alone group
Statistical Analysis 4: Comparison: Part A: mRNA-1345 + Afluria® Quadrivalent vs Part A: Afluria® Quadrivalent + Placebo; Influenza B Phuket Antibody; Test type: Non-Inferiority — Lower bound of the 95% CI of geometric mean ratio (GMR) >0.667, using a noninferiority margin of 1.5; GMR = 0.909, 95% CI 2-sided [0.809 to 1.020] — mRNA-1345+Afluria group at Day 29 compared with the GMT of anti-HA Ab in the Afluria alone group

37. Primary Outcome: Part B: Number of Participants With Solicited Local and Systemic ARs Within 7 Days After Day 1 Injection
Description: Solicited ARs were collected in an eDiary. Local ARs: injection site pain, erythema (redness), swelling/induration (hardness); and axillary (underarm) swelling or tenderness ipsilateral to the side of injection. Systemic ARs: fever, headache, fatigue, myalgia, arthralgia, nausea/vomiting, and chills. Note, not all solicited ARs were considered AEs. Investigator reviewed whether the solicited AR was also to be recorded as an AE. A Summary of SAEs and nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Within 7 days after Day 1 injection
Population: Solicited Safety Set included all randomized participants who received any study intervention and contributed any solicited ARs data from the time of study injection on Day 1 through the following 6 days. Participants were included in the treatment arm corresponding to the study drug they actually received. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo | Part B: mRNA-1273.214 + Placebo + Placebo
Number analyzed (Participants) | 553 | 557 | 556
Participants | 358 | 394 | 361

38. Primary Outcome: Part B: Number of Participants With Solicited Local and Systemic ARs Within 7 Days After Day 29 Injection
Description: as for outcome 37
Time Frame: Within 7 days after Day 29 injection
Population: Part B Solicited Safety Set Day 29 Injection consisted of all randomized participants who received any study injection on Day 29 and contributed any solicited ARs. Participants were included in the treatment arm corresponding to the study drug they actually received. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo | Part B: mRNA-1273.214 + Placebo + Placebo
Number analyzed (Participants) | 522 | 532 | 528
Participants | 265 | 147 | 148

39. Primary Outcome: Part B: Number of Participants With Unsolicited AEs After Day 1 Injection
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Any abnormal laboratory test result (hematology, clinical chemistry, or PT/PTT) or other safety assessment (for example, electrocardiogram, radiological scan, vital sign measurement), including one that worsened from baseline and was considered clinically significant in the medical and scientific judgment of the Investigator was recorded as an AE. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Day 1 through Day 28 (28 days after Day 1 injection)
Population: Safety Set Day 1 injection included all randomized participants who received any study intervention. Participants were included in the treatment arm corresponding to the study drug they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo | Part B: mRNA-1273.214 + Placebo + Placebo
Number analyzed (Participants) | 554 | 562 | 560
Participants | 41 | 54 | 44

40. Primary Outcome: Part B: Number of Participants With Unsolicited AEs After Day 29 Injection
Description: as for outcome 32
Time Frame: Day 29 through Day 57 (28 days after Day 29 injection)
Population: Safety Set Day 29 injection included all randomized participants who received any study intervention. Participants were included in the treatment arm corresponding to the study drug they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo | Part B: mRNA-1273.214 + Placebo + Placebo
Number analyzed (Participants) | 530 | 535 | 536
Participants | 31 | 25 | 26

41. Primary Outcome: Part B: Number of Participants With MAAEs, SAEs, AESIs, and AEs Leading to Withdrawal
Description: as for outcome 33
Time Frame: Day 1 through Day 211
Population: Safety Set included all randomized participants who received any study intervention. Participants were included in the treatment arm corresponding to the study drug they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo | Part B: mRNA-1273.214 + Placebo + Placebo
Number analyzed (Participants) | 554 | 562 | 560
Participants
  MAAEs | 109 | 107 | 97
  SAEs | 18 | 13 | 10
  AESIs | 5 | 2 | 7
  AEs Leading to Withdrawal | 1 | 0 | 0

42. Primary Outcome: Part B: GMT of Serum RSV-A at Day 29
Description: Antibody values reported as below LLOQ were replaced by 0.5*LLOQ. Values greater than the upper limit of quantification (ULOQ) were replaced by the ULOQ. LLOQ was 13 IU/mL and ULOQ was 259061 IU/mL for RSV-A. As prespecified, only arms where participants received mRNA-1345 are presented for this outcome measure.
Time Frame: Day 29
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo
Number analyzed (Participants) | 508 | 506
IU/mL | 19071.03 [17130.14 to 21231.84] | 15171.23 [13626.94 to 16890.53]
Statistical Analysis 1: Comparison: Part B: mRNA-1345 + Placebo + mRNA-1273.214 vs Part B: mRNA-1345 + mRNA-1273.214 + Placebo; Test type: Non-Inferiority — Lower bound of the 95% CI of ratio of the GMT (GMR) >0.667, using a noninferiority margin of 1.5; GMR = 0.796, 95% CI 2-sided [0.702 to 0.901] — mRNA-1345+mRNA-1273.214 compared to mRNA-1345 alone

43. Primary Outcome: Part B: Percentage of Participants With Seroresponse for RSV-A Neutralizing Abs From Baseline to Day 29
Description: as for outcome 2
Time Frame: Baseline to Day 29
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo
Number analyzed (Participants) | 508 | 506
percentage of participants | 75.4 [71.4 to 79.1] | 70.9 [66.8 to 74.9]
Statistical Analysis 1: Comparison: Part B: mRNA-1345 + Placebo + mRNA-1273.214 vs Part B: mRNA-1345 + mRNA-1273.214 + Placebo; Test type: Non-Inferiority — Lower bound of the 95% CI of the SRR difference >-10%, using noninferiority margin of 10%; Difference = -4.4, 95% CI 2-sided [-9.9 to 1.0] — mRNA-1345+mRNA-1273.214 compared to mRNA-1345 alone

44. Primary Outcome: Part B: Geometric Mean Concentration (GMC) of Serum Ab Level, as Measured by Neutralization Assay for SARS-Cov-2 at Day 29
Description: The model-based GM titer was estimated on ANCOVA model. SARS-CoV-2 variants included Wuhan-Hu-1 and B.1.1.529. Antibody values reported as below LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ were replaced by the ULOQ. LLOQ was 10 arbitrary units (AU)/milliliters (mL) and ULOQ was 111433 AU/mL for Wuhan-Hu-1. LLOQ was 8 and ULOQ was B.1.1.529 for B1.1.529. As prespecified, only arms where participants received mRNA-1273.214 are presented for this outcome measure.
Time Frame: Day 29
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: AU/mL
Arm/Group | Part B: mRNA-1345 + mRNA-1273.214 + Placebo | Part B: mRNA-1273.214 + Placebo + Placebo
Number analyzed (Participants) | 513 | 519
AU/mL
  Wuhan-Hu-1: number analyzed (Participants) | 501 | 512
  Wuhan-Hu-1 | 9881.69 [9097.35 to 10733.66] | 10300.49 [9490.13 to 11180.04]
  B.1.1.529 | 2353.15 [2115.26 to 2617.80] | 2342.87 [2107.26 to 2604.82]
Statistical Analysis 1: Comparison: Part B: mRNA-1345 + mRNA-1273.214 + Placebo vs Part B: mRNA-1273.214 + Placebo + Placebo; GMR for Wuhan-Hu-1; Test type: Non-Inferiority — Lower bound of the 95% CI of ratio of the GMT (GMR) >0.667, using a noninferiority margin of 1.5; GMR = 0.959, 95% CI 2-sided [0.872 to 1.056] — mRNA-1345+mRNA-1273.214 compared to mRNA-1273.214 alone
Statistical Analysis 2: Comparison: Part B: mRNA-1345 + mRNA-1273.214 + Placebo vs Part B: mRNA-1273.214 + Placebo + Placebo; GMR for B.1.1.529; Test type: Non-Inferiority — Lower bound of the 95% CI of ratio of the GMT (GMR) >0.667, using a noninferiority margin of 1.5; GMR = 1.004, 95% CI 2-sided [0.888 to 1.137] — mRNA-1345+mRNA-1273.214 compared to mRNA-1273.214 alone

45. Primary Outcome: Part B: Percentage of Participants With Seroresponse for SARS-Cov-2 NAbs From Baseline to Day 29
Description: Seroresponse was defined as ≥4 × LLOQ if baseline was <LLOQ or 4-fold or greater increase from baseline if baseline was ≥LLOQ. mRNA-As prespecified, only arms where participants received mRNA-1273.214 are presented for this outcome measure.
Time Frame: Baseline to Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part B: mRNA-1345 + mRNA-1273.214 + Placebo | Part B: mRNA-1273.214 + Placebo + Placebo
Number analyzed (Participants) | 513 | 519
percentage of participants
  Wuhan-Hu-1: number analyzed (Participants) | 501 | 512
  Wuhan-Hu-1 | 52.7 [48.2 to 57.1] | 52.5 [48.1 to 56.9]
  B.1.1.529 | 68.4 [64.2 to 72.4] | 69.4 [65.2 to 73.3]
Statistical Analysis 1: Comparison: Part B: mRNA-1345 + mRNA-1273.214 + Placebo vs Part B: mRNA-1273.214 + Placebo + Placebo; SRR difference for Wuhan-Hu-1; Test type: Non-Inferiority — Lower bound of the 95% CI of the SRR difference >-10%, using noninferiority margin of 10%; Difference = 0.2, 95% CI 2-sided [-6.0 to 6.3] — mRNA-1345+mRNA-1273.214 compared to mRNA-1273.214 alone
Statistical Analysis 2: Comparison: Part B: mRNA-1345 + mRNA-1273.214 + Placebo vs Part B: mRNA-1273.214 + Placebo + Placebo; SRR difference for B.1.1.529; Test type: Non-Inferiority — Lower bound of the 95% CI of the SRR difference >-10%, using noninferiority margin of 10%; Difference = -0.9, 95% CI 2-sided [-6.6 to 4.7] — mRNA-1345+mRNA-1273.214 compared to mRNA-1273.214 alone

46. Primary Outcome: Part C: Number of Participants With Solicited Local and Systemic Within 7 Days After Revaccination Day 1
Description: Solicited ARs were collected in an electronic eDiary. Local ARs: injection site pain, erythema (redness), swelling/induration (hardness); and axillary (underarm) swelling or tenderness ipsilateral to the side of injection. Systemic ARs: fever, headache, fatigue, myalgia, arthralgia, nausea/vomiting, and chills. Note, not all solicited ARs were considered AEs. Investigator reviewed whether the solicited AR was also to be recorded as an AE. A Summary of SAEs and nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Within 7 days after Day 1 revaccination
Population: Solicited Safety Set included all participants who received revaccination with mRNA-1345 and contributed any solicited AR data. Participants were included in the treatment arm corresponding to the study drug they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- Part C: mRNA-1345 Revaccincation: Overall participants who received a single mRNA-1345 primary vaccination on Day 1 in Part B and then received revaccination with a single mRNA-1345 injection at least 12 months later (but not longer than 15 months) (Revaccination Day 1).
Arm/Group | Part C: mRNA-1345 Revaccincation
Number analyzed (Participants) | 543
Participants | 338

47. Primary Outcome: Part C: Number of Participants With Unsolicited AEs Within 28 Days After Revaccination Day 1
Description: as for outcome 39
Time Frame: Revaccination Day 1 through Day 28 (28 days after revaccination Day 1)
Population: Safety Set included all participants who received any revaccination with mRNA-1345. Participants were included in the treatment arm corresponding to the study drug they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: mRNA-1345 Revaccincation
Number analyzed (Participants) | 543
Participants | 31

48. Primary Outcome: Part C: Number of Participants With MAAEs
Description: A MAAE is an AE that leads to an unscheduled visit to a healthcare practitioner.
Time Frame: Revaccination Day 1 through Day 181
Population: as for outcome 47
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: mRNA-1345 Revaccincation
Number analyzed (Participants) | 543
Participants | 105

49. Primary Outcome: Part C: Number of Participants With SAEs, AESIs, and AEs Leading to Withdrawal
Description: An SAE was defined as any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability, was a congenital anomaly/birth defect, or was an important medical event. An AESI is an AE (serious or nonserious) of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor are required. A summary of SAEs and all nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: Revaccination Day 1 through Day 361
Population: as for outcome 47
Measure: Count of Participants; unit: Participants
Arm/Group | Part C: mRNA-1345 Revaccincation
Number analyzed (Participants) | 543
Participants
  SAEs | 28
  AESIs | 2
  AEs Leading to Withdrawal | 5

50. Primary Outcome: Part C: GMT of Serum RSV-A and RSV-B NAbs mRNA-1345 Revaccination Day 29 Compared to Primary Vaccination Day 29
Description: Antibody values reported as below LLOQ were replaced by 0.5*LLOQ. Values greater than the ULOQ were replaced by the ULOQ. LLOQ was 13 IU/mL and ULOQ was 259061 IU/mL for RSV-A. LLOQ was 10 IU/mL and ULOQ was 112476 IU/mL for RSV-B.
  mRNA-1345 Revaccination Day 29 and mRNA-1345 primary vaccination Day 29 (received in Part B) are presented.
Time Frame: Primary Vaccination Day 29 to Revaccination Day 29
Population: PP Set: participants received mRNA-1345 revaccination, had prerevaccination and at least 1 postinjection assessment of immunogenicity after revaccination, complied with immunogenicity testing schedule, and had no major protocol derivations. 'Overall number of participants analyzed' = participants evaluable for this endpoint. 'Number analyzed' = participants evaluable for specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Part C: mRNA-1345 Primary Vaccination | Part C: mRNA-1345 Revaccincation
Number analyzed (Participants) | 524 | 525
IU/mL
  RSV-A: number analyzed (Participants) | 519 | 525
  RSV-A | 18190.30 [16467.13 to 20093.79] | 19649.18 [18017.92 to 21428.12]
  RSV-B | 6746.41 [6136.32 to 7417.16] | 6123.47 [5599.77 to 6696.14]
Statistical Analysis 1: Comparison: Part C: mRNA-1345 Primary Vaccination vs Part C: mRNA-1345 Revaccincation; GMR of RSV-A. GMR was calculated by back transforming the mean of paired difference of antibody levels on the logarithmic scale between revaccination Day 29 and primary vaccination Day 29; Test type: Non-Inferiority — Lower bound of the 95% CI of ratio of the GMT (GMR) >0.667, using a noninferiority margin of 1.5; GMR = 1.077, 95% CI 2-sided [0.995 to 1.166] — The 95% CI for the GMR is based on t-distribution of the log-transformed values then back transformed to the original scale for presentation
Statistical Analysis 2: Comparison: Part C: mRNA-1345 Primary Vaccination vs Part C: mRNA-1345 Revaccincation; GMR of RSV-B. GMR was calculated by back transforming the mean of paired difference of antibody levels on the logarithmic scale between revaccination Day 29 and primary vaccination Day 29; Test type: Non-Inferiority — Lower bound of the 95% CI of ratio of the GMT (GMR) >0.667, using a noninferiority margin of 1.5; GMR = 0.909, 95% CI 2-sided [0.839 to 0.984] — [estimate comment as in outcome 50, analysis 1]

51. Other Pre Specified Outcome: Number of Deaths During the Study
Description: A death that occurred during the study or that came to the attention of the investigator during the study was reported to the Sponsor, whether or not it was considered related to study drug. The investigator assessed causality (that is, whether there is a reasonable possibility that the study drug caused the death). The relationship was characterized using the following classifications: Not related: There was not a reasonable possibility of a relationship to the study drug. The temporal sequence of the death relative to administration of the study drug was not reasonable and/or the death was more likely explained by a cause other than the study drug. Related: There was a reasonable possibility of a relationship to the study drug. There was evidence of exposure to the study drug. The temporal sequence of the death relative to the administration of the study drug was reasonable. The death was more likely explained by the study drug than by another cause.
Time Frame: Up to Day 181 for Part A, up to Day 211 for Part B, and up to Day 361 for Part C
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: mRNA-1345 + Placebo | Part A: mRNA-1345 + Afluria® Quadrivalent | Part A: Afluria® Quadrivalent + Placebo | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo | Part B: mRNA-1273.214 + Placebo + Placebo | Part C: mRNA-1345 Revaccination
Number analyzed (Participants) | 249 | 690 | 692 | 560 | 564 | 562 | 543
Participants
  Deaths | 0 | 3 | 1 | 1 | 0 | 0 | 3
  Deaths related to study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality and serious adverse events were collected throughout the entire period of the study (up to Day 181 for Part A, up to Day 211 for Part B, and up to Day 361 for Part C). Other (not including serious) adverse events were collected for 28 days after the vaccination unless they met the criteria for AESIs, MAAEs or AEs led to discontinuation.
Description: The serious and other (not including serious) adverse events were based on the safety set which consisted of all randomized participants who received the study drug. Adverse event data were collected during the study visit by the investigator. A participant may experience the same event both as SAE and non-SAE.
Groups:
- Part A: mRNA-1345 + Afluria Quadrivalent: Participants received a single injection each of mRNA-1345 and Afluria® quadrivalent, administered IM on Day 1.
- Part A: Afluria Quadrivalent + Placebo: Participants received a single injection each of Afluria® quadrivalent and placebo, administered IM on Day 1.
- Part C: Revaccination: Participants received mRNA-1345 primary vaccination in Part B and opted to receive revaccination in Part C. Participants received a single mRNA-1345 injection at least 12 months (but not longer than 15 months) after primary vaccination.
Arm/Group | Part A: mRNA-1345 + Placebo | Part A: mRNA-1345 + Afluria Quadrivalent | Part A: Afluria Quadrivalent + Placebo | Part B: mRNA-1345 + Placebo + mRNA-1273.214 | Part B: mRNA-1345 + mRNA-1273.214 + Placebo | Part B: mRNA-1273.214 + Placebo + Placebo | Part C: Revaccination
All-Cause Mortality (participants affected / at risk) | 0/249 | 3/690 | 1/692 | 1/560 | 0/564 | 0/562 | 3/543
Serious Adverse Events (participants affected / at risk) | 4/249 | 28/685 | 24/689 | 18/554 | 13/562 | 10/560 | 28/543
Other Adverse Events (participants affected / at risk) | 0/249 | 0/685 | 0/689 | 0/554 | 0/562 | 0/560 | 0/543
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: mRNA-1345 + Placebo (N=249) | Part A: mRNA-1345 + Afluria Quadrivalent (N=685) | Part A: Afluria Quadrivalent + Placebo (N=689) | Part B: mRNA-1345 + Placebo + mRNA-1273.214 (N=554) | Part B: mRNA-1345 + mRNA-1273.214 + Placebo (N=562) | Part B: mRNA-1273.214 + Placebo + Placebo (N=560) | Part C: Revaccination (N=543)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metapneumovirus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — A participant in the Part C: Revaccination group experienced a fatal SAE of septic shock considered unrelated to study drug by the investigator.
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — A participant in the Part A: mRNA-1345 + Afluria Quadrivalent group experienced a fatal SAE of gastric cancer considered unrelated to study drug by the investigator.
Hepatic cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuroendocrine tumour of the rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Triple negative breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — A participant in the Part C: Revaccination group experienced a fatal SAE of diabetic ketoacidosis considered unrelated to study drug by the investigator.
Acute psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium tremens (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subdural effusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — A participant in the Part C: Revaccination group experienced a fatal SAE of cardiac arrest considered unrelated to study drug by the investigator.
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — A participant in the Part A: Afluria Quadrivalent + Placebo group experienced a fatal SAE of cardiac failure considered unrelated to study drug by the investigator.
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Superficial vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venous occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Necrotising oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — A participant in the Part A: mRNA-1345 + Afluria Quadrivalent group and a participant in the Part B: mRNA-1345 + Placebo + mRNA-1273.214 group had SAEs of death considered unrelated to study drug by the investigator.
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — A participant in the Part A: mRNA-1345 + Afluria Quadrivalent group experienced a fatal SAE of subdural hematoma (secondary to a fall) considered unrelated to study drug by the investigator.
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT05330975/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT05330975/SAP_001.pdf